CLINICAL TRIAL: NCT06066346
Title: Talquetamab Consolidation After BCMA CART Cell Therapy for Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of Talquetamab for People With Multiple Myeloma Who Have Received BCMA CAR T-Cell Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Janssen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-072
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
Keywords: Talquetamab; BCMA CAR T-Cell Therapy; 23-072
MeSH Terms: conditions — Multiple Myeloma | interventions — talquetamab

STUDY DESIGN:
Intervention Model Description: Single arm phase II trial
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Talquetamab (Experimental): Subcutaneous Talquetamab
  Interventions: Drug: Talquetamab

INTERVENTIONS:
Drug: Talquetamab — Talquetamab will be administered SC until disease progression

SUMMARY:
The researchers are doing this study to find out whether talquetamab is an effective treatment after BCMA CAR Tcell therapy for people with relapsed or refractory multiple myeloma. All participants in this study will have already received the BCMA CAR T-cell therapy ide-cel for their disease.

ELIGIBILITY:
Inclusion Criteria:

* Patient with multiple myeloma who has received prior treatment with an IMID, PI, and a CD38 monoclonal antibody
* Received treatment with an FDA approved BCMA CART cell therapy ide-cel within 1-3 months prior to enrollment
* Serum monoclonal protein < 0.5 gm/dL; 24-hour urine monoclonal protein < 200 mg; and serum involved free light chains < 10 mg/dL
* No evidence of disease progression based on IMWG criteria
* ≥18 years of age at the time of signing informed consent.
* ECOG performance status of 0 or 1
* Recovered to Grade 1 or baseline of any non-hematologic toxicities due to prior treatments, excluding Grade 2 neuropathy and Grade 2 alopecia.
* No evidence of ongoing, any grade cytokine release syndrome or immune effector cell mediated neurotoxicity
* No additional myeloma therapies after the CART cell therapy
* Absolute neutrophil count (ANC) ≥ 1,000/mm^3 without growth factor support for 7 days for G-CSF or GM-CSF and for 14 days for pegylated GCSF prior to the laboratory test.
* Platelet count ≥ 75,000/mm^3 (without platelet transfusion or thrombopoietin receptor agonist use in the previous 7 before the laboratory test). Platelets ≥ 50,000/mm^3 is acceptable if the counts prior lymphodepleting chemotherapy for the preceding CAR T cell therapy was < 75,000.
* Hemoglobin ≥ 8 g/dL (without red blood cell transfusion support or erythropoietin use within 7 days of the laboratory test).
* Creatinine Clearance (CrCl)/estimated glomerular filtration rate (eGFR) ≥ 30 mL/min, measured by 24 hour urine assessment or estimated by CKD-EPI2021.
* Oxygen saturation ≥ 92% on room air
* Hepatic Function:

  * Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x upper limit of normal (ULN)
  * Serum total bilirubin ≤ 2 x ULN; except in participants with congenital bilirubinemia, such as Gilbert syndrome (in which case direct bilirubin ≤1.5 x ULN is required).
* International ratio (INR) or partial thromboplastin time (PTT) < 1.5 x ULN
* Cardiac Function: left ventricular ejection fraction ≥ 45% by echocardiogram (ECHO) or multigated acquisition scan (MUGA).
* Willing and able to adhere to the study visit schedule and other protocol requirements
* Female patients of childbearing potential (FCBP) must:

  * Have a negative highly-sensitive serum β-human chorionic gonadotropin (β-hCG) pregnancy test (<5 IU/mL) at screening and a negative urine or serum pregnancy test within 24 hours before the first dose of study drug.
  * Practicing a highly effective, preferably user-independent method of contraception (failure rate of <1% per year when used consistently and correctly) and agrees to remain on a highly effective method while receiving study drug and until 100 days after last dose.
  * Agree to pregnancy testing (serum or urine) within 100 days after the last study drug administration.
  * Agree to use an additional contraceptive method in addition to the requirements listed above
  * Agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for at least 100 days after the last dose of study drug.
  * Agree to abstain from breastfeeding from screening through at least 6 months after the last dose of talquetamab
* Male patients must:

  * Agree to wear a condom when engaging in any activity that allows for passage of ejaculate to another person, during the study and for 100 days after the last dose of study drug. Male subjects should also be advised of the benefit for a female partner to use a highly effective method of contraception as a condom may break or leak.
  * Men must agree not to donate sperm for the purpose of reproduction during the study and for at least 100 days after receiving the last dose of study drug.
* Must sign an ICF (or their legally acceptable representative must sign) indicating that the participant understands the purpose of, and procedures required for, the study and is willing to participate in the study.

Exclusion Criteria:

* Prior or concurrent exposure to any of the following in the specified time frame prior to enrollment:

  * Received any prior GRPRC5D-directed therapy
  * T-cell redirection therapy (for example, antibody therapy or BiTE's) within 3 months
  * Investigational vaccine other than SARS CoV-2 vaccine approved/ in use under emergency approval within 4 weeks
  * Live, attenuated vaccine within 4 weeks.
  * Monoclonal antibody therapy within 21 days (with the exception of COVID monoclonal antibodies)
  * Cytotoxic therapy within 21 days
  * PI therapy within 14 days
  * IMiD agent therapy within 14 days
  * Radiotherapy within 14 days or focal radiation within 7 days
  * Major surgery (as defined by the investigator) within 14 days
  * Plasmapheresis within 14 days
* Received either of the following:

  * An allogeneic SCT within 6 months before the first dose of study treatment. Participants who received an allogeneic transplant must be off all immunosuppressive medications during the 6 weeks before the start of study treatment administration without signs of graft-versus-host disease.
  * An autologous SCT within 12 weeks before the start of study treatment administration
* A maximum cumulative dose of corticosteroids of ≥ 140 mg of prednisone or equivalent within 14-day period before the first dose of study drug (does not include pretreatment medications).
* Prior organ transplant requiring systemic immunosuppressive therapy
* History of ≥ Grade 2 hemorrhage within 30 days of enrollment
* Patient requiring ongoing treatment with chronic, therapeutic dosing of anticoagulants (e.g., Warfarin, low molecular weight heparin, Factor Xa inhibitors) can be enrolled with approval of the PI.
* History or presence of clinically relevant CNS pathology such as epilepsy, seizure, paresis, aphasia, stroke, subarachnoid hemorrhage or other CNS bleed, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis. Additionally, any patients with meningeal or CNS involvement of MM will be excluded.
* Having concurrent Waldenstrom's macroglobulinemia, POEMS (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes), active plasma cell leukemia, or clinically significant amyloidosis
* History of Class III or IV congestive heart failure (CHF) or severe nonischemic cardiomyopathy, unstable or poorly controlled angina, myocardial infarction, or hemodynamically significant ventricular arrhythmia within the previous 6 months prior to enrollment
* Active clinically significant autoimmune disease, defined as a history of requiring systemic immunosuppressive therapy and at ongoing risk for potential disease exacerbation. Patients with a history of autoimmune thyroid disease, asthma, or limited skin manifestations are potentially eligible. Patients with a history of acute or chronic GVHD are potentially eligible if on minimal immunosuppressants as defined previously.
* Seropositive for human immunodeficiency virus (HIV-1). Acute hepatitis A. Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Subjects with resolved infection (ie, subjects who are HBsAg negative with antibodies to total hepatitis B core antigen [Anti-HBc] with or without the presence of hepatitis B surface antibodies [Anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of HBVDNA levels. Those who are PCR positive will be excluded. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (Anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR. Active hepatitis C infection as measured by positive hepatitis C virus (HCV)-RNA testing. Subjects with a history of Hepatitis C virus antibody positivity must undergo HCV-RNA testing
* Prior malignancies except resected basal cell carcinoma or treated carcinoma in situ. Cancer treated with curative intent less than 5 years prior to enrollment will not be allowed unless approved by the PI. Cancer treated with curative intent greater than 5 years prior to enrollment is allowed.
* Myelodysplastic syndrome or active malignancies (ie, progressing or requiring treatment change in the last 24 months) other than relapsed/refractory multiple myeloma. The only allowed exceptions are:

  * Non-muscle invasive bladder cancer treated within the last 24 months that is considered completely cured
  * Skin cancer (non-melanoma or melanoma) treated within the last 24 months that is considered completely cured.
  * Noninvasive cervical cancer treated within the last 24 months that is considered completely cured
  * Localized prostate cancer (N0M0):
  * With a Gleason score of ≤6, treated within the last 24 months, or untreated and under surveillance
  * With a Gleason score of 3+4 that has been treated >6 months prior to full study screening and considered to have a very low risk of recurrence
  * History of localized prostate cancer and receiving androgen deprivation therapy and considered to have a very low risk of recurrence.
  * Breast cancer: adequately treated lobular carcinoma in situ or ductal carcinoma in situ, or history of localized breast cancer and receiving antihormonal agents and considered to have a very low risk of recurrence
  * Other malignancy that is considered cured with minimal risk of recurrence.
* Female patients who are breastfeeding or who intend to become pregnant during participation in the study or until 100 days after the last dose of therapy.
* Participant plans to father a child while enrolled in this study or within 100 days after the last dose of study treatment.
* Known allergy or hypersensitivity to any of the study medications, their analogues, or excipients in the various formulations of any agent.
* Serious medical of psychiatric illness likely to interfere with participation on this clinical study
* Uncontrolled bacterial, viral or fungal infections (currently taking medication and with progression or no clinical improvement) at time of enrollment.
* Acute diffuse infiltrative pulmonary disease requiring home oxygen therapy
* Unwilling or unable to provide informed consent
* Unable or unwilling to return to the center for treatment and follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | up to 2 years
  ORR is defined as the proportion of participants who have a partial response (PR) or better according to the international myeloma working group (IMWG) criteria.

SECONDARY OUTCOMES:
Rate of sustained Minimal Residual Disease (MRD) | 2 years
  negativity in the bone marrow (defined as MRD negativity determined at least 12 months apart).

CONTACTS AND LOCATIONS:
Overall Officials: Sham Mailankody, MBBS, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm